CLINICAL TRIAL: NCT07370805
Title: Prospective Clinical Study and Exploration of 18F-FAPI PET/CT Imaging in Lung Cancers
Brief Title: 18F-FAPI PET in Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: FirstZhejiangU-FAPI-Lung Ca
Record Dates: First submitted 2025-12-25; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer (Diagnosis)
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- FAPI-Lung-ca: 18F FAPI PET scans
  Interventions: Diagnostic Test: 18F-FAPI PET

INTERVENTIONS:
Diagnostic Test: 18F-FAPI PET — 1、Patients clinically suspected or confirmed with lung cancer are required to complete conventional imaging examinations (CT/MR or FDG PET) and undergo ¹⁸F-FAPI PET/CT.

SUMMARY:
This study aims to evaluate the diagnostic efficacy and prognostic value of 18F-FAPI PET/CT in lung cancer.

DETAILED DESCRIPTION:
1. Patients clinically suspected or confirmed with lung cancer are required to complete conventional imaging examinations (CT/MR or FDG PET) and undergo ¹⁸F-FAPI PET/CT.
2. Conduct a detailed inquiry into the patient's medical history to clarify symptoms, signs, and prior medical history (e.g., tumor history, surgical history, biopsy history, radiotherapy history, chemotherapy history, family history, allergy history, etc.), as well as relevant laboratory tests and previous imaging findings (including plain radiography, ultrasound, CT, MRI, 18F-FDG PET/CT, PET/MR, etc.).
3. For follow-up coordination, you are required to regularly provide your clinical data (e.g., treatment plans, disease progression, etc.) as per the study requirements. This collaboration is essential for completing long-term follow-up, including monitoring the subject's condition, imaging findings, pathological results (such as tumor grading and Ki-67 index), and patient treatment outcomes, to collect prognostic information.
4. ¹⁸F-FAPI PET/CT and conventional imaging examinations (e.g., CT/MR) were completed prior to enrollment. After enrollment in this study, subjects were not required to undergo additional imaging or laboratory tests, only requiring follow-up without intervention to the clinical treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Lung Cancer
2. With 18F FAPI PET scan

Exclusion Criteria:

1. Concurrent presence of other active malignant tumors or a history of other
2. malignant tumors within the past 5 years;
3. Severe uncontrollable diseases or active infections;
4. Ineligible participants for project informed consent；
5. Pregnant and lactating women.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | through study completion, an average of 1.5 year
  Sensitivity, specificity, positive and negative predictive value of 18F-FAPI PET Imaging in lung cancer.

SECONDARY OUTCOMES:
Standard uptake value （SUV）of tumor | through study completion, 3-4 years
  This measure evaluates the association between baseline 18F-FAPI PET parameters (e.g., SUVmax, SUVmean).
Metabolic tumor volume (c) and total lesion glycolysis (TLG) of tumor | through study completion, 3-4 years
  This measure evaluates the association between baseline 18F-FAPI PET parameters (MTV in cm3, TLG in cm3*SUV）
Prognostic Value of Baseline 18F-FAPI PET for Progression-Free Survival (PFS) in High-Risk Patients | through study completion, 3-4 years
  PFS will be defined as the time from diagnosis to disease progression or relapse, assessed using the Kaplan-Meier method and Cox proportional hazards model.（PFS in months）

CONTACTS AND LOCATIONS:
Overall Officials: Donghe Chen, MD, Study Director — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-11-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT07370805/Prot_ICF_000.pdf